CLINICAL TRIAL: NCT04059419
Title: PARQUE 70+ Studying Sleep Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Marcia Uchoa Rezende, Full Professor in Orthopedics and Traumatology, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cappesq 04019418.7.0000.0068
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Osteoarthritis; Sleep Disorder
Keywords: Osteoarthritis; Quality of Life; Sleep disorder
MeSH Terms: conditions — Osteoarthritis; Sleep Wake Disorders | interventions — Health Services for the Aged

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): 30 Patients will participate in two days of lectures two-months apart on the subject of knee OA, but will also come to the hospital at months 1, 3 and 5 after the first class to consult about nutritional habits to be improved; at months 4 and 6 to participate in a group therapy session with the psychologists, 7 sessions with the physical therapy team followed by 7 sessions with the physical educators team (once a week/4 weeks and once every two weeks, three times).
  Interventions: Behavioral: PARQVE Program
- Control (Active Comparator): Should remain under geriatric care after randomization.
  Interventions: Behavioral: Geriatric Care

INTERVENTIONS:
Behavioral: PARQVE Program — Two days of lectures about knee OA, come to the hospital at months 1, 3 and 5 after the first class to consult about nutritional habits to be improved, participate in a group therapy session with the psychologists and sessions with the physical educators.
  Arms: Experimental
Behavioral: Geriatric Care — Remain under geriatric care as usual
  Arms: Control

SUMMARY:
The emerging Brazilian population is accompanied by the emergence of patients in an age group, including osteoarthritis. Osteoarthritis (OA) is one of the most prevalent musculoskeletal diseases, affecting 4% of the Brazilian population. By 2050, 30% of Brazil's population is over 60 years old. This has a higher degree of elderly with morbades as unbass on the association, such as osteoarthritis. Proper management of OA involves educational program, multidisciplinary team care and therapeutic maneuvers with weight loss and maintenance of mobility. Insomnia is the most frequent sleep disorder in the elderly and its execution almost always harms young women. Sleep quality is interfered with fatigue and pain exacerbation in people with OA, ie a sleep approach should be diagnosed in patients with comorbidity. In addition, chronic patients usually have insomnia and pressure in the use of opioids, sedatives and antidepressants, pointing to insomnia and mood swings for polypharmacy. To evaluate a quality of sleep as an intervention of the PARQVE 70+ Project. Prospective, case-control study. Patients over 70 years old treated at a geriatric outpatient clinic with eye or polyarticular osteoarthesis and clinical OA treatment indicator will be allocated and matched in two groups of 30 elderly. Patients underwent Pittsburgh Sleep Quality Index questionnaires and the Epworth Scale before the study began, 3 and 6 months after PARQVE interventions and number of analysts, and compared those who did not perform an intervention. The study aims to improve sleep quality, decrease pain, reduce quality and decrease daytime sleepiness in elderly with OA.

DETAILED DESCRIPTION:
The growing Brazilian population aging is accompanied by the emergence of common diseases in this age group, including osteoarthritis. Osteoarthritis (OA) is the most prevalent musculoskeletal disease, affecting 4% of the Brazilian population. There is important morbidity which progressively leads to chronic use of drugs harmful to this age group, such as anti-inflammatory drugs, increasing the risk of complications and pharmacological interactions. In addition to culminating with disabling functional impairment, osteoarthritis may progress, leading to the need for arthroplasty. Obesity and longevity are important risk factors for osteoarthritis, and both are very prevalent in Brazil.

2010 IBGE census progressions suggest a growing population increase, with 13% of the Brazilian population in 2018. By 2050, 30% of Brazil's population will be over 60 years old. This reflects a gradual increase in the elderly with common morbidities in this age group, such as osteoarthritis. Proper management of OA involves an educational program, multidisciplinary team care, and therapeutic measures aimed at weight loss and maintaining mobility.

Insomnia is the most frequent sleep disorder in the elderly and its prevalence almost doubles compared to young adults. In addition to aging, other factors such as the presence of clinical comorbidities, including OA, psychiatric disorders, primary sleep disorders and poor habits (poor sleep hygiene) contribute to this prevalence. During the aging process, in addition to increased nighttime awakenings and increased total waking time at night, there is a reduction in time spent in the deepest stages of sleep, which may be compromised in the presence of pain.

Sleep quality is affected by severe fatigue and pain exacerbation in people with OA, ie the sleep approach should always be considered in patients with such comorbidity. In addition to OA, patients with chronic pain usually have insomnia and depression, increasing the use of opioids, sedatives and antidepressants, indicating insomnia and mood changes contributing factors to polypharmacy.

A systematic review of chronic OA pain and spinal pain suggests that interventions such as cognitive behavioral therapy and sleep hygiene have good repercussions in people with OA.

The study of sleep improvement can facilitate the elderly's quality of life, decrease pain and reduce polypharmacy. This study aims to evaluate the improvement of sleep quality and decrease of daytime sleepiness in elderly with OA.

ELIGIBILITY:
Inclusion Criteria:

* Classified as Kelgreen and Lawrence grades I to III (K-L), ie any degree of gonarthritis without obliteration of the joint space;
* Indication of clinical treatment of OA;
* Patients without moderate to advanced dementia syndrome;
* Patients without neuropsychiatric diseases whose symptoms may impair the assimilation of the given guidelines.

Exclusion Criteria:

* Missing interventions and not performing the tasks determined by professionals;
* Patients with low family support;
* Prescription in the last three months, during the study, some type of hypnotic or sleep inducing medication, which may interfere with the study analysis.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate changes in the quality of sleep after the multiprofessional intervention | 6 months
  Answer questionnaires about sleep disorders - Ranges Min: 0 Better - Max: 24 Worse

SECONDARY OUTCOMES:
Change of the insomnia severity index | Baseline, 3 months and 6 months
  Answer insomnia severity index - Ranges Min: 0 Better - Max: 24 Worse
Change of the Epworth Sleepiness Scale | Baseline, 3 months and 6 months
  Answer Epworth Sleepiness Scale - Ranges Min: 0 Better - Max: 24 Worse
Change of the subjective complaint of perception of sleep | Baseline, 3 months and 6 months
  Answer the subjective complaint of perception of sleep - Ranges Min: 0 Better - Max: 24 Worse
Change in the amount of pain medication | Baseline, 3 months and 6 months
  Take notes day by day amount of medication

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme Ocampos, MD, Principal Investigator — University of São Paulo General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hawker GA, Badley EM, Borkhoff CM, Croxford R, Davis AM, Dunn S, Gignac MA, Jaglal SB, Kreder HJ, Sale JE. Which patients are most likely to benefit from total joint arthroplasty? Arthritis Rheum. 2013 May;65(5):1243-52. doi: 10.1002/art.37901. PMID 23459843
- [Background] Ferreira MC, Oliveira JCP, Zidan FF, Franciozi CEDS, Luzo MVM, Abdalla RJ. Total knee and hip arthroplasty: the reality of assistance in Brazilian public health care. Rev Bras Ortop. 2018 Jun 8;53(4):432-440. doi: 10.1016/j.rboe.2018.05.002. eCollection 2018 Jul-Aug. PMID 30027075
- [Background] Rezende MU, Frucchi R, Pailo AF, Campos GC, Pasqualin T, Hissadomi MI. PARQVE: PROJECT ARTHRITIS RECOVERING QUALITY OF LIFE THROUGH EDUCATION: TWO-YEAR RESULTS. Acta Ortop Bras. 2017 Jan-Feb;25(1):18-24. doi: 10.1590/1413-785220172501165604. PMID 28642645
- [Background] Bliwise DL. Sleep in normal aging and dementia. Sleep. 1993 Jan;16(1):40-81. doi: 10.1093/sleep/16.1.40. No abstract available. PMID 8456235
- [Background] Wolkove N, Elkholy O, Baltzan M, Palayew M. Sleep and aging: 1. Sleep disorders commonly found in older people. CMAJ. 2007 Apr 24;176(9):1299-304. doi: 10.1503/cmaj.060792. PMID 17452665
- [Background] Fu K, Makovey J, Metcalf B, Bennell KL, Zhang Y, Asher R, Robbins SR, Deveza LA, Cistulli PA, Hunter DJ. Sleep Quality and Fatigue Are Associated with Pain Exacerbations of Hip Osteoarthritis: An Internet-based Case-crossover Study. J Rheumatol. 2019 Nov;46(11):1524-1530. doi: 10.3899/jrheum.181406. Epub 2019 Apr 1. PMID 30936279
- [Background] Liu M, McCurry SM, Belza B, Buchanan DT, Dobra A, Von Korff M, Vitiello MV. Effects of Pain, Insomnia, and Depression on Psychoactive Medication Supply in Older Adults With Osteoarthritis. Med Care. 2018 Dec;56(12):1024-1031. doi: 10.1097/MLR.0000000000000982. PMID 30256279
- [Background] Ho KKN, Ferreira PH, Pinheiro MB, Aquino Silva D, Miller CB, Grunstein R, Simic M. Sleep interventions for osteoarthritis and spinal pain: a systematic review and meta-analysis of randomized controlled trials. Osteoarthritis Cartilage. 2019 Feb;27(2):196-218. doi: 10.1016/j.joca.2018.09.014. Epub 2018 Oct 18. PMID 30342087